CLINICAL TRIAL: NCT03912272
Title: Effectiveness of Long-term Low-frequency High-Intensity Interval Training (HIIT) to Improve Body Adiposity and Liver Fat in Adults With Central Obesity: A Randomized Controlled Trial
Brief Title: 12-Month Once-a-week HIIT Improves Body Adiposity and Liver Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Parco M. Siu, PhD, Associate Professor and Division Head, Division of Kinesiology, School of Public Health, Li Ka Shing Faculty of Medicine, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RF-9835-NAFLD-001
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Central Obesity
Keywords: Long-Term Low-Frequency High-Intensity Interval Training; Non-Alcoholic Fatty Liver Disease; Central Obesity; Body Adiposity; Liver Fat
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity, Abdominal; Fatty Liver | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Control (Placebo Comparator): Subjects in the usual care control group will receive a health education program. This program includes 12-month twice-a-month sessions (70 minutes each session) for obesity-related health briefing, dietary caloric restriction advice, and lifestyle counseling/consultation. The class will be conducted in small group setting (4-8 participants each group). The same health information will be delivered to the subjects in the HIIT group throughout the 12-month intervention period. Subjects will be asked to attend >70% of the classes.
  Interventions: Behavioral: Usual Care Control
- High-intensity Interval Training Group (Experimental): HIIT will be prescribed once weekly under the supervision of certified athletics coaches for 12 months. HIIT training will be performed in a small group setting (4-8 participants each group) in laboratories. In each session, subjects will run for four 4-minute intervals at 85%-95% of the peak heart rate (HRpeak) with a 3-minute active recovery at 50%-70% of the HRpeak between each interval. A 5-minute jog at an intensity of 70% of the HRpeak will be included for warm-up and cool-down before and after, respectively. Subjects will be asked to attend >70% of the classes.
  Interventions: Behavioral: High-intensity Interval Training

INTERVENTIONS:
Behavioral: High-intensity Interval Training — In the high-intensity interval training group, subjects will receive respective prescribed exercise once a week.
  Arms: High-intensity Interval Training Group
Behavioral: Usual Care Control — In the usual care control group, obesity-related health briefing, dietary caloric restriction advice, and lifestyle counseling/consultation will be provided.
  Arms: Usual Care Control

SUMMARY:
Obesity and non-alcoholic fatty liver disease (NAFLD) are two related growing epidemics that are becoming pressing public health concerns. High-intensity interval training (HIIT) is a promising cost-effective and time-efficient exercise modality for managing obesity and NAFLD. However, patients with obesity and NAFLD are generally inactive and unfit, and might feel intimidated by the frequency of the prescribed HIIT (conventionally three times weekly). Previous HIIT studies, mostly over 2-4 month periods, showed that the participants could accomplish this exercise frequency under a controlled laboratory environment, but the long-term adherence and sustainability, especially in a field setting, remains uncertain. The situation is more unclear if we also consider those individuals who refused to participate possibly because of their overwhelming perceptions or low self-efficacy toward HIIT. Thus, logically, HIIT at a lower frequency would be practical and more suitable for patients with obesity and NAFLD, but the minimum exercise frequency required to improve health, especially in the long-term, is unknown. This proposed study aims to examine the effectiveness of long-term low-frequency HIIT for improving body adiposity and liver fat in centrally obese adults. The premise of this proposal is supported by recent findings that HIIT performed once a week could improve cardiorespiratory fitness, blood pressure, cardiac morphology, metabolic capacity, muscle power, and lean mass. This study will provide evidence for the benefits of long-term low-frequency HIIT with a follow-up period to assess its effectiveness, safety, adherence, and sustainability. We expect this intervention will enhance the practical suitability of HIIT in inactive obese adults and will provide evidence for low-frequency HIIT as a new exercise option in the management of obesity and NAFLD.

ELIGIBILITY:
Inclusion Criteria:

1. Cantonese, Mandarin or English speaking,
2. Aged 18-60,
3. Central obesity, defined as BMI ≥25 (obesity classification adopted by the Hong Kong Government) with waist circumference of ≥90 cm for men and ≥80 cm for women (abdominal obesity according to the International Diabetes Federation's Chinese ethnic-specific criterion),
4. Willing to initiate lifestyle modification but not pharmacologic or surgical means for treating obesity.

Exclusion criteria:

1. ≥150 minutes moderate-intensity exercise or ≥75 minutes vigorous exercise weekly,
2. Regular HIIT (≥1 weekly) in the past six months,
3. Medical history of cardiovascular disease, chronic pulmonary or kidney disease, heart failure, cancer, and liver disease except for NAFLD,
4. Somatic conditions that limit exercise participation (e.g., limb loss),
5. Impaired mobility due to chronic diseases (e.g., chronic arthritis/osteoarthritis, neurological, musculoskeletal and autoimmune diseases),
6. Daily smoking habit,
7. Excess alcohol consumption (daily ≥30 g of alcohol for men and ≥20 g for women) in the past six months
8. Surgery, therapy or medication for obesity or weight loss in the past 6 months (e.g., gastric bypass, gastric band, sleeve gastrectomy, gastric reduction duodenal switch, and dietitian-prescribed dietary program).
9. During the study period, subjects identified with major physical changes that would considerably affect their body composition and weight (e.g., anorexia nervosa, bulimia nervosa, and prolonged gastrointestinal and digestive disorders) will be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-09-07 (Actual); Study Completion 2024-09-07 (Actual)

PRIMARY OUTCOMES:
Liver Fat | Change from baseline amount of intrahepatic triglycerides content at 12 months
  Intrahepatic triglycerides will be examined by 1H-MR spectroscopy in a 3×3×3 cm voxel using a 1.5-Tesla scanner (SIGNA™ Explorer - 60cm, General Electric Healthcare) housed at the MR imaging unit of HKU core facility. A trained MRI radiographer will operate the machine, position the subjects and analyze the results. NAFLD will be defined as >5% intrahepatic triglycerides assessed by 1H-MR spectroscopy.
Body Adiposity | Change from baseline amount of body fat mass at 12 months
  Total body fat mass will be determined using a full body dual-energy X-ray absorptiometry (DXA) scanner (Explorer S/N 91075, Hologic Inc., Waltham, USA). A trained technician will operate the DXA machine, position the subjects and analyze the results. The typical coefficients of variation of the DXA scanner for each body compartment from duplicate analyses are 0.4% for lean mass, 1.4% for fat mass and 1.0% for bone mass
Liver Fat | Change from baseline amount of intrahepatic triglycerides content at 24 months
  Intrahepatic triglycerides will be examined by 1H-MR spectroscopy in a 3×3×3 cm voxel using a 1.5-Tesla scanner (SIGNA™ Explorer - 60cm, General Electric Healthcare) housed at the MR imaging unit of HKU core facility. A trained MRI radiographer will operate the machine, position the subjects and analyze the results. NAFLD will be defined as >5% intrahepatic triglycerides assessed by 1H-MR spectroscopy.
Body Adiposity | Change from baseline amount of body fat mass at 24 months
  Total body fat mass will be determined using a full body dual-energy X-ray absorptiometry (DXA) scanner (Explorer S/N 91075, Hologic Inc., Waltham, USA). A trained technician will operate the DXA machine, position the subjects and analyze the results. The typical coefficients of variation of the DXA scanner for each body compartment from duplicate analyses are 0.4% for lean mass, 1.4% for fat mass and 1.0% for bone mass

SECONDARY OUTCOMES:
Visceral Adiposity | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up
  Abdominal visceral fat will be measured using a three-point Dixon sequence using a 1.5-Tesla scanner (SIGNA™ Explorer - 60cm, General Electric Healthcare) housed at the MR imaging unit of HKU core facility. A trained MRI radiographer will operate the machine, position the subjects and analyze the results. The abdominal visceral fat between the thoracic diaphragm and the upper bORDER of the first sacral vertebra will be manually marked on each MRI transverse image to calculate the volume of abdominal visceral fat.
Subcutaneous Adiposity | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up
  Subcutaneous fat will be measured using a three-point Dixon sequence using 1.5-Tesla scanner (SIGNA™ Explorer - 60cm, General Electric Healthcare) housed at the MR imaging unit of HKU core facility. A trained MRI radiographer will operate the machine, position the subjects and analyze the results. The abdominal subcutaneous fat between the thoracic diaphragm and the upper border of the first sacral vertebra will be manually marked on each MRI transverse
Body Mass Index | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up
  A calibrated electronic digital weighing scale (UC321, A&D Medical) with a capacity from 0.05kg to 150kg (± 0.05kg accuracy) will be used to weigh the subjects. A stadiometer (Holtain Ltd., UK) with 200 cm limit and ± 0.01 cm accuracy will be used to measure body height. The BMI will be calculated from the body weight and height.
Waist Circumference | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up
  Waist circumference will be measured on bare skin midway between the lowest rib and the superior border of the iliac crest using an inelastic measuring tape to the nearest 0.1 cm. Measurement will be performed at the end of normal expiration.
Hip Circumference | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up
  Hip circumference will be be taken on bare skin around the widest portion of the buttocks using an inelastic measuring tape to the nearest 0.1 cm and the tape should be placed parallel to the floor.
VO2max | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up
  VO2max test will be conducted using a calibrated motor-driven treadmill (LE500C, Jaeger, Germany) by continuous metabolic VO2 measurement using a Cosmed K5 portable telemetric gas analysis system. The test will be performed using a ramp protocol where the speed will be constant and the incline will be increased by 2% every second minute until VO2max is reached. Capillary blood will be obtained before and immediately after the test for the blood lactate analysis. The highest value of VO2 which meets one of the following criteria will be considered as the VO2max: 1) plateau of VO2 with increasing intensity, 2) respiratory exchange ratio (RER) ≥1.05, and 3) post-exercise blood lactate exceeding 8 mmol/L.
Blood Pressure | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up
  Subjects will abstain from consuming caffeine and alcohol at least 10 hours prior to the assessment. After 10 minutes rest in the seated position, blood pressure will be measured on the right arm using a blood pressure monitor (M3 Vital Signs Monitor, EDAN). Systolic and diastolic blood pressure and mean arterial pressure will be obtained over the brachial artery region with the arm supported at the heart level using an appropriately sized cuff. Measurements will be repeated after 10 minutes and the average of two separate measurements will be recorded for the analysis.
Lean Mass | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up
  Total body lean mass will be determined by using DXA scan.
Bone Mineral Density | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up
  Bone mineral density will be determined by using DXA scan.
Fasting glucose | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up
  Subjects will fast overnight for 10 hours. Subjects will sit in a quiet environment for 15 minutes prior to blood collection. Venous blood will be drawn from an antecubital vein in the forearm by a certified phlebotomist and sent to an accredited medical laboratory to measure the level of fasting glucose.
Insulin | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up
  Subjects will fast overnight for 10 hours. Subjects will sit in a quiet environment for 15 minutes prior to blood collection. Venous blood will be drawn from an antecubital vein in the forearm by a certified phlebotomist and sent to an accredited medical laboratory to measure the level of insulin.
HbA1c | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up
  Subjects will fast overnight for 10 hours. Subjects will sit in a quiet environment for 15 minutes prior to blood collection. Venous blood will be drawn from an antecubital vein in the forearm by a certified phlebotomist and sent to an accredited medical laboratory to measure the level of HbA1c.
Alanine aminotransferase ALT | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up
  Subjects will fast overnight for 10 hours. Subjects will sit in a quiet environment for 15 minutes prior to blood collection. Venous blood will be drawn from an antecubital vein in the forearm by a certified phlebotomist and sent to an accredited medical laboratory to measure the level of ALT.
Aspartate aminotransferase AST | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up
  Subjects will fast overnight for 10 hours. Subjects will sit in a quiet environment for 15 minutes prior to blood collection. Venous blood will be drawn from an antecubital vein in the forearm by a certified phlebotomist and sent to an accredited medical laboratory to measure the level of AST.
LDL cholesterol | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up
  Subjects will fast overnight for 10 hours. Subjects will sit in a quiet environment for 15 minutes prior to blood collection. Venous blood will be drawn from an antecubital vein in the forearm by a certified phlebotomist and sent to an accredited medical laboratory to measure the level of LDL cholesterol.
HDL cholesterol | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up.
  Subjects will fast overnight for 10 hours. Subjects will sit in a quiet environment for 15 minutes prior to blood collection. Venous blood will be drawn from an antecubital vein in the forearm by a certified phlebotomist and sent to an accredited medical laboratory to measure the level of HDL cholesterol.
Total cholesterol | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up.
  Subjects will fast overnight for 10 hours. Subjects will sit in a quiet environment for 15 minutes prior to blood collection. Venous blood will be drawn from an antecubital vein in the forearm by a certified phlebotomist and sent to an accredited medical laboratory to measure the level of total cholesterol.
Triglycerides | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up.
  Subjects will fast overnight for 10 hours. Subjects will sit in a quiet environment for 15 minutes prior to blood collection. Venous blood will be drawn from an antecubital vein in the forearm by a certified phlebotomist and sent to an accredited medical laboratory to measure the level of triglycerides.
Class adherence | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up
  Class attendance will be recorded to indicate adherence to HIIT intervention. Subjects will be encouraged to achieve >70% class attendance over the year.
Dropout rate | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up
  The reasons for dropout will be ascertained and reported.
Dose-response relationship between attendance and other outcome variables | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up
  Secondary analysis will be performed based on the attendance rate to examine the dose-response relationship between HIIT and the other outcome variables.
Quality of Life measured by Short Form-12 | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up
  The validated Chinese version Standard SF-12 Health Survey will be used to measure health-related quality of life. This 12-item questionnaire assesses physical functioning, emotional and mental health, bodily pain, general health, vitality and social functioning. A higher overall score indicates better quality of life.
Mental Health measured by the Hospital Anxiety and Depression Scale (HADS) | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up
  The Hospital Anxiety and Depression Scale (HADS) will also be used to evaluate the severity of depression and anxiety. This 7-item questionnaire has an overall score ranging from 0 to 21 (with subscales for both anxiety and depression). A higher score indicates more severe symptoms.
Anxiety level measured by Generalized Anxiety Disorder-7 (GAD-7) | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up
  Generalized Anxiety Disorder-7 (GAD-7) will also be used to measure the anxiety level of the subjects. This 7-item questionnaire has an overall score ranging from 0 to 21. A higher score indicates more severe symptoms.
Depression level measured by Patient Health Questionnaire-9 (PHQ-9) | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up
  Patient Health Questionnaire-9 (PHQ-9) will also be used to measure the depression level of the subjects. This 10-item questionnaire has an overall score ranging from 0 to 30. A higher score indicates more severe symptoms.
Sleep Quality | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up
  Pittsburgh Sleep Quality Index (PSQI) will be used to measure the subjective sleep quality of the subjects. The score of this scale ranges from 0 to 21. Higher score indicates worse subjective sleep quality.
Adverse Events | The adverse events will be recorded during the one-year intervention period
  Adverse events will be closely monitored through regular surveys by the athletics coaches and research personnel, and by voluntary reports from the subjects. The incidence rate in both usual care control group and HIIT group will be calculated as incidence rate = number of adverse events in each group / number of participants in each group.
Medication usage | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up
  The number of participants in each group using dyslipidemic and hypertensive medications will be recorded, including e.g., drug name, type, dose and weekly frequency).
Habitual Physical Activity | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up
  Habitual physical activity will be measured by International Physical Activity Questionnaire (IPAQ) and 7-day actigraph. Subjects will wear the actigraph at the hip region for 24 hours over 8 consecutive days. The first day will be a trial and not be included into the analysis.
Dietary Intake | All assessments will be repeated at 12 months post-intervention and at 24 months at the follow-up
  The dietary intake will be measured by 3-day weighed food record and analyzed by Food Processor, ESHA. A food ingestion report will be generated by the software, including total calories intake, proportion of major macro nutrients.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Fai Parco Siu, PhD, Principal Investigator — Li Ka Shing Faculty of Medicine, The University of Hong Kong
Locations (1):
- Li Ka Shing Faculty of Medicine, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The data of individual participants that underlie the results reported in this trial, after de-identification including text, tables, figures, and appendices, as well as study protocol and statistical analysis plan, will be shared after 3 months of study publication. Data will be shared with researchers who provide a methodologically sound proposal for academic purposes. Proposals should be directed to pmsiu@hku.hk to gain access and for data request, a data-access agreement needs to be signed.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 3 years following the publication of the article
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal for academic purposes. Proposals should be directed to pmsiu@hku.hk to gain access and for data request, a data-access agreement needs to be signed.

REFERENCES:
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Siu PM, Yu AP, Benzie IF, Woo J. Effects of 1-year yoga on cardiovascular risk factors in middle-aged and older adults with metabolic syndrome: a randomized trial. Diabetol Metab Syndr. 2015 Apr 30;7:40. doi: 10.1186/s13098-015-0034-3. eCollection 2015. PMID 26000038
- [Background] Siu PM. Efficacy of Tai Chi training to alleviate insomnia in older adults. Proceeding of The 6th International Conference on Nutrition and Physical Activity (NAPA 2015), Taipei, Taiwan 2015;p.59
- [Background] Siu PM, Yu AP, Yu DS, Hui SS, Woo J. Effectiveness of Tai Chi training to alleviate metabolic syndrome in abdominal obese older adults: A randomized controlled trial.
- [Background] Siu PM, Yu AP, Yu DS, Hui SS, Woo J. Effects of Tai Chi Exercise on Cardiometabolic Health and Muscle Content. Proceeding of the 3rd Asian Conference for Frailty and Sarcopenia, Seoul, Korea 2017
- [Background] Ramos JS, Dalleck LC, Borrani F, Beetham KS, Mielke GI, Dias KA, Wallen MP, Keating SE, Fassett RG, Coombes JS. High-intensity interval training and cardiac autonomic control in individuals with metabolic syndrome: A randomised trial. Int J Cardiol. 2017 Oct 15;245:245-252. doi: 10.1016/j.ijcard.2017.07.063. Epub 2017 Jul 21. PMID 28747269
- [Background] Ramos JS, Dalleck LC, Borrani F, Beetham KS, Wallen MP, Mallard AR, Clark B, Gomersall S, Keating SE, Fassett RG, Coombes JS. Low-Volume High-Intensity Interval Training Is Sufficient to Ameliorate the Severity of Metabolic Syndrome. Metab Syndr Relat Disord. 2017 Sep;15(7):319-328. doi: 10.1089/met.2017.0042. Epub 2017 Jun 22. PMID 28846513
- [Background] Ramos JS, Dalleck LC, Borrani F, Mallard AR, Clark B, Keating SE, Fassett RG, Coombes JS. The effect of different volumes of high-intensity interval training on proinsulin in participants with the metabolic syndrome: a randomised trial. Diabetologia. 2016 Nov;59(11):2308-2320. doi: 10.1007/s00125-016-4064-7. Epub 2016 Aug 1. PMID 27480182
- [Background] Ramos JS, Dalleck LC, Ramos MV, Borrani F, Roberts L, Gomersall S, Beetham KS, Dias KA, Keating SE, Fassett RG, Sharman JE, Coombes JS. 12 min/week of high-intensity interval training reduces aortic reservoir pressure in individuals with metabolic syndrome: a randomized trial. J Hypertens. 2016 Oct;34(10):1977-87. doi: 10.1097/HJH.0000000000001034. PMID 27467767
- [Background] Siu PM, Chin EC, Wong SH, Fong DY, Chan DK, Ngai HH, Lee CH, Yung PS. Low-frequency high-intensity interval training (HIIT) improves cardiorespiratory fitness and body composition in overweight adults. Med Sci Sports Exerc 2018:abstract submitted to the 65th American College of Sports Medicine (ACSM) Annual Meeting.
- [Derived] Chin EC, Leung CK, Yu DJ, Yu AP, Bernal JK, Lai CW, Chan DKC, Ngai HH, Yung PSH, Lee CH, Fong DY, Keating SE, Coombes JS, Siu PM. Effects of one-year once-weekly high-intensity interval training on body adiposity and liver fat in adults with central obesity: Study protocol for a randomized controlled trial. J Exerc Sci Fit. 2022 Apr;20(2):161-171. doi: 10.1016/j.jesf.2022.03.003. Epub 2022 Mar 14. PMID 35401766